CLINICAL TRIAL: NCT00753818
Title: Developmental Effects of Infant Formula Supplemented With LCPUFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Other Study IDs: 3370-2(-4); NCT00222157 (obsolete NCT alias)
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: Cognitive Development; Growth
Keywords: infant formula; visual development

ARMS (4):
- 1 (Experimental)
  Interventions: Other: DHA and ARA
- 2 (Experimental)
  Interventions: Other: DHA and ARA
- 3 (Experimental)
  Interventions: Other: DHA and ARA
- 4 (Other): Control
  Interventions: Other: Control

INTERVENTIONS:
Other: DHA and ARA — various levels of DHA and ARA
  Arms: 1; 2; 3
Other: Control
  Arms: 4

SUMMARY:
The purpose of this study is to compare the effects on visual development, growth, cognitive development, tolerance, and blood chemistry parameters in term infants fed one of four study formulas containing various levels of DHA and ARA.

ELIGIBILITY:
Inclusion Criteria:

* healthy, term, formula fed infants from 1-5 days of age

Exclusion Criteria:

* history of disease that effects normal growth and development
* breast fed, or formula intolerance

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child

PRIMARY OUTCOMES:
visual development

SECONDARY OUTCOMES:
Cognitive development

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Kansas Medical Center, Kansas City, Kansas
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Derived] Liao K, McCandliss BD, Carlson SE, Colombo J, Shaddy DJ, Kerling EH, Lepping RJ, Sittiprapaporn W, Cheatham CL, Gustafson KM. Event-related potential differences in children supplemented with long-chain polyunsaturated fatty acids during infancy. Dev Sci. 2017 Sep;20(5):10.1111/desc.12455. doi: 10.1111/desc.12455. Epub 2016 Oct 16. PMID 27747986
- [Derived] Drover JR, Felius J, Hoffman DR, Castaneda YS, Garfield S, Wheaton DH, Birch EE. A randomized trial of DHA intake during infancy: school readiness and receptive vocabulary at 2-3.5 years of age. Early Hum Dev. 2012 Nov;88(11):885-91. doi: 10.1016/j.earlhumdev.2012.07.007. Epub 2012 Jul 25. PMID 22835597
- [Derived] Birch EE, Carlson SE, Hoffman DR, Fitzgerald-Gustafson KM, Fu VL, Drover JR, Castaneda YS, Minns L, Wheaton DK, Mundy D, Marunycz J, Diersen-Schade DA. The DIAMOND (DHA Intake And Measurement Of Neural Development) Study: a double-masked, randomized controlled clinical trial of the maturation of infant visual acuity as a function of the dietary level of docosahexaenoic acid. Am J Clin Nutr. 2010 Apr;91(4):848-59. doi: 10.3945/ajcn.2009.28557. Epub 2010 Feb 3. PMID 20130095